CLINICAL TRIAL: NCT02917083
Title: Phase I Study of Relapsed CD30 Expressing Lymphoma Treated With CD30 CAR T Cells (RELY-30)
Brief Title: CD30 CAR T Cells, Relapsed CD30 Expressing Lymphoma (RELY-30)
Acronym: RELY-30
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-37966, RELY-30; RELY-30 (Other: Center for Cell and Gene Therapy)
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin Lymphoma
Keywords: chimeric antigen receptors; immunotherapy; CAR T-cells; lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD30.CAR T Cells (Experimental): Each patient will receive one infusion of CAR modified T cells. Unless post autologous transplant, patients will receive lymphodepleting chemotherapy as three daily doses of cyclophosphamide (Cy: 500mg/m2/day) together with fludarabine (Flu:30mg/m2/day) from 48 hours to 2 weeks before T cell infusion. Clofarabine (20 mg/m2/day) may be substituted for fludarabine.
  Interventions: Genetic: CAR T Cells

INTERVENTIONS:
Genetic: CAR T Cells — Three dose levels will be evaluated based on safety data from our current study of CD30 CAR T cells. Cohorts of three to six patients will be enrolled at each dose level. Each patient will receive one infusion of CAR modified T cells according to the following dosing schedule:
  Dose Level One: 2x10^7 cells/m2. Dose Level Two: 1x10^8 cells/m2. Dose Level Three: 2x10^8 cells/m2.
  Other Names: CD30.CAR T Cells

SUMMARY:
The subject has a type of lymph gland cancer called Lymphoma.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with germs. Both antibodies and T cells have been used to treat patients with cancers; they both have shown promise, but have not been strong enough to cure most patients. Investigators hope that both will work better together.

Investigators have found from previous research that they can put a new gene into T cells that will make them recognize cancer cells and kill them. They now want to test whether these genetically modified T cells given after chemotherapy will be more effective at killing cancer cells.

The gene that will be put into the T cells makes an antibody called anti-CD30. This antibody sticks to lymphoma cells because of a substance on the outside of the cells called CD30. Anti-CD30 antibodies have been used to treat people with lymphoma, but have not been strong enough to cure most patients.

For this study, the anti-CD30 antibody has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD30 chimeric receptor-activated T cells (CD30.CAR T cells) seem to kill some of the tumor, but they don't last very long and so their chances of fighting the cancer are unknown.

Several studies suggest that the infused T cells need room to be able to multiply and grow to accomplish their functions, and that this may not happen if there are too many other T cells in circulation. Because of that, doctors may use chemotherapy drugs to decrease the level of circulating T cells prior to the CD30.CAR T cells infusion. This is called "lymphodepletion"

CD30.CAR T cells have previously been studied in lymphoma patients.

DETAILED DESCRIPTION:
To prepare the CD30.CAR T cells, research staff will take some blood from the subject. This would be drawn as two separate blood collections.

Alternatively, if the subject's blood counts are low, staff may collect the cells needed to prepare T cells by a pheresis procedure. This procedure will involve placing a needle in both arms, collecting the cells over 3 to 6 hours during which the subject will be required to lie relatively still.

After the T cells have been collected, some of them will be activated stimulating them with antibodies and will then be infected with a retroviral vector (a special virus that can carries a new gene into cells) containing a new gene called anti-CD30 that will make an antibody to lymphoma cells. The trained cells are called CD30.CAR T cells. Then, the cells will be tested to make sure that they kill lymphoma cells that express the CD30 antigen and not normal cells.

The cells generated will be frozen and stored to give back to the subject.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest doses (1 of 3 different levels) of CD30.CAR T Cells. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 3 dose levels are studied. If the side effects are too severe, the dose will be lowered or the T cell infusions will be stopped. The risks of harm and discomfort from the study treatment may bear some relationship to the dose level. The potential for direct benefit, if any, may also vary with the dose level.

Subjects will be given one injection of CD30.CAR T cells. The injection will be on Day 0. The subject may be given a dose of Benadryl and Tylenol before the injection of T cells to minimize any possible allergic reaction. The injection will take 1-10 minutes. The subject will be monitored in the clinic after each injection for at least 3 hours.

At the discretion of the study doctor, if the subject has stable disease (the lymphoma did not grow) or there is a reduction in the size of the lymphoma on imaging studies at week 8 after the T-cell infusion or on subsequent evaluations, then the subject can receive up to six additional doses of the T cells at 8 to 12 weeks intervals. After each T cell injection, the subject will be monitored as described above.

To learn more about the way the CD30.CAR T cells are working and how long they last in the body, extra blood will be drawn. On the day that the subject receives the cells, blood will be taken before the cells are given and several hours afterwards. For patients receiving lymphodepletion chemotherapy blood will also be collected prior to the start of chemotherapy. Other blood will be drawn at 1 week, 2 weeks, 3 weeks (optional), 4 weeks, 6 weeks and 8 weeks, every 3 months for 1 year, every 6 months for 4 years, then yearly for a total of 15 years.

ELIGIBILITY:
PROCUREMENT Inclusion Criteria:

1. Diagnosis of relapsed/refractory HL or NHL.
2. CD30 positive tumor as assayed in a CLIA certified pathology laboratory (result can be pending at this time)
3. Hgb ≥ 7.0 (may be a transfused value)
4. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.
5. Karnofsky or Lansky score of > 60%

TREATMENT Inclusion Criteria:

1. Diagnosis of relapsed/refractory HL or NHL.
2. CD30-positive tumor as assayed in a CLIA certified pathology laboratory.
3. Age 16 to 75 for the first three patients on a dose level; thereafter, if no DLT, patients aged 12 to 75 can be treated on that dose level.
4. Bilirubin 1.5 times or less than the upper limit of normal.
5. AST 3 times or less than the upper limit of normal.
6. Estimated GFR > 70 mL/min.
7. Pulse oximetry of > 90% on room air
8. EKG shows no significant arrhythmias
9. Karnofsky or Lansky score of > 60%.
10. Available autologous T cells with greater than or equal to 15% expression of CD30CAR determined by flow-cytometry.
11. Recovered from all acute non-hematologic toxic effects of all prior chemotherapy.
12. Adequate pulmonary function with FEV1, FVC and DLCO (or DLCO/VA, as clinically appropriate) greater than or equal to 50% of expected corrected for hemoglobin.
13. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
14. Informed consent explained to, understood by and signed by patient or guardian.

PROCUREMENT Exclusion Criteria:

1. Active infection with HIV or HTLV (can be pending at this time).
2. Active bacterial, fungal or viral infection.

TREATMENT Exclusion Criteria:

1. Currently receiving any investigational agents or received any tumor vaccines within the previous six weeks.
2. Received anti-CD30 antibody-based therapy within the previous 4 weeks.
3. Subjects with rapidly progressive disease, defined as kinetic failure to previous chemotherapy.
4. Bulky disease (defined as a 10 cm or greater mass or mediastinal disease with a transverse diameter exceeding 33% of the transthoracic diameter).
5. History of hypersensitivity reactions to murine protein-containing products.
6. Pregnant or lactating.
7. Tumor in a location where enlargement could cause airway obstruction.
8. Current use of systemic corticosteroids at a dose equivalent to 0.5 mg/kg/day of prednisone or higher.
9. Active hemorrhagic cystitis.
10. Active bacterial, viral or fungal infection.
11. Symptomatic cardiac disease (NYHA Class III or IV disease).

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2040-02 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-Limiting Toxicities (DLT) | 6 weeks
  Each treated patient will be followed for 6 weeks post the T-cell infusion for the evaluation of DLTs.

SECONDARY OUTCOMES:
Median Number of T cells transduced with the vector | 15 years
  The investigators will monitor the persistence of these infused cells by measuring the level of the transgene by both phenotypic and molecular analyses.
Overall Response Rate | 8 weeks
  Although response is not the primary endpoint of this trial, investigators will summarize tumor response by calculating overall response rates along with exact 95% binomial confidence intervals.
Mean Number of T cells transduced with the vector | 15 years
  The investigators will monitor the persistence of these infused cells by measuring the level of the transgene by both phenotypic and molecular analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos CA, Grover NS, Beaven AW, Lulla PD, Wu MF, Ivanova A, Wang T, Shea TC, Rooney CM, Dittus C, Park SI, Gee AP, Eldridge PW, McKay KL, Mehta B, Cheng CJ, Buchanan FB, Grilley BJ, Morrison K, Brenner MK, Serody JS, Dotti G, Heslop HE, Savoldo B. Anti-CD30 CAR-T Cell Therapy in Relapsed and Refractory Hodgkin Lymphoma. J Clin Oncol. 2020 Nov 10;38(32):3794-3804. doi: 10.1200/JCO.20.01342. Epub 2020 Jul 23. PMID 32701411